CLINICAL TRIAL: NCT05625698
Title: Axillary Lymph Node Identification Before Neoadjuvant Chemotherapy Using MagTrace (Superparamagnetic Iron Oxide Nanoparticles, SPIO) and Magseed, in Clinically Node Negative and Node Positive Patients: a Feasibility Study.
Brief Title: Premarking of Axillary Nodes Before Start of Neoadjuvant Chemotherapy Using Magnetic Approach
Acronym: SENTINEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Professor, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SUGBG-2021002
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy, sentinel node, axillary clearance
MeSH Terms: conditions — Breast Neoplasms | interventions — ferric oxide

STUDY DESIGN:
Intervention Model Description: This is a feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MagTrace only (Other): Cohort 1: Clinically node negative patients undergoing neoadjuvant chemotherapy. This cN0-group will receive MagTrace injections before start of neoadjuvant chemotherapy followed standard routine technetium-99 injections after neoadjuvant chemotherapy to facilitate surgery. Nodes containing Magtrace will be detected by finding the magnetic signals using the SentiMag probe. No other interventions during chemotherapy treatments
  Interventions: Drug: MagTrace only
- MagTrace and Magseed (Other): Cohort 2: Clinically node positive patients undergoing neoadjuvant chemotherapy. This N+ group will receive MagTrace injection in the breast to mark sentinel nodes and Magseed will be inserted into the index metastatic node before the start of neoadjuatnt chemotherapy followed by standard routine technetium-99 injections after neoadjuvant chemotherapy to facilitate surgery. Nodes containing Magtrace / Magseed will be detected by finding the magnetic signals using the SentiMag probe. No other interventions during chemotherapy treatments
  Interventions: Combination Product: MagTrace and Magseed

INTERVENTIONS:
Drug: MagTrace only — see information in arm descriptions
  Other Names: SPIO
  Arms: MagTrace only
Combination Product: MagTrace and Magseed — see information in arm descriptions
  Other Names: SPIO
  Arms: MagTrace and Magseed

SUMMARY:
Breast cancer is one of the commonest types of cancers in females. Treatments include surgery followed by anti-estrogen therapy, radiotherapy and chemotherapy. During breast surgery, the surgeon removes the cancer from the breast and lymph nodes (glands) from the armpit.

Historically, all armpit lymph nodes were surgically removed but this approach is associated long term problems of arm swelling. In more recent times, an increasingly more selective approach is used to treat the armpit nodes. In the presence of cancer spreads in the nodes, an axillary clearance surgery is done otherwise, only the first node(s) also called sentinel node(s) that drain fluids from the cancer, is surgically removed. The identification of nodes using the latter approach is helped by injecting a tracer in the breast and via the lymphatic channels, the tracer is then concentrated in the sentinel nodes.

Over recent years, neoadjuvant (preoperative) chemotherapy is being increasingly used to treat breast cancers. This treatment approach can lead up to a large of number of complete cancer response. This in turn can cause difficulties in locating the breast cancer / armpit nodes during surgery after the chemotherapy.

New developments like superparamagnetic iron oxide nanoparticles (SPIO or MagTrace®) has been used as an alternate liquid tracer to mark sentinel nodes to facilitate armpit surgery. In addition, small magnetic clip called Magseed® has also been developed which can be inserted into the relevant lymph nodes thereby marking their anatomical position to facilitate surgery. Both MagTrace and Magseed can be used to pre-mark the cancer and armpit nodes before the start of neoadjuvant chemotherapy. In theory, premarking armpit nodes using a magnetic approach is associated with better surgical accuracy in the armpit but there is limited supporting data.

Therefore, this study aims to investigate the feasibility of premarking armpit nodes, with or without cancer spread, using magtrace and magseed respectively before patients undergo neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is one of the commonest types of cancers in females. Treatments include surgery followed by anti-estrogen therapy (tablet form), radiotherapy (radiation) and chemotherapy (intravenous / tablet form). During breast surgery, the surgeon removes the cancer from the breast and lymph nodes (glands) from the armpit.

Historically, all armpit lymph nodes (clearance) were removed irrespective of the stage of armpit disease which can lead to over-treatment and unnecessary long term arm lymphoedema (swelling). However, the modern approach has become more selective. If there are cancer spread in the nodes at diagnosis, a clearance operation is carried out otherwise only the first node(s) that the cancer spreads to, is removed. The latter procedure is called sentinel node biopsy and it is usually done by injecting a radioactive liquid tracer near the breast cancer. The tracer is then drained via the breast lymphatic channels and concentrated in the relevant armpit nodes where it can be detected by using a detector probe during surgery.

In recent years, there are increasing uses of preoperative (neoadjuvant, NACT) chemotherapy in certain breast cancer subtypes with good cancer response. In up to 70% of cases, the treated cancer had disappeared both, in the breast and armpit, after NACT. Consequently, it can be difficult to locate and surgically remove these nodes in the armpits even with the usual injection of tracer after NACT. These difficulties are due to the damage of lymphatic channels in the breast by NACT and become fibrotic. Therefore, the tracer injected after NACT will no longer be drained correctly to mark the correct nodes in the armpit as the lymphatic channels are altered. In turn, this can lead to wrong sentinel nodes being removed from the armpit, which then can cause inaccurate planning for further treatments.

Over recent times, superparamagnetic iron oxide nanoparticles (SPIO or MagTrace®) has been used as an alternate liquid tracer to mark sentinel nodes to facilitate armpit surgery. In addition, small magnetic clip called Magseed® has also been developed. Magseed® can be directly inserted into the relevant lymph nodes thereby marking their anatomical position to facilitate surgery. Both MagTrace and Magseed are longer lasting materials in the body than the radioactive technetium. Therefore, these new techniques give rise to an opportunity to premark the armpit nodes before the damage to lymphatic channels (with MagTrace) and before the cancer in the nodes disappear (with magseed), after NACT. In theory, premarking armpit nodes using a magnetic approach is associated with better surgical accuracy in the armpit but there is limited supporting data.

Therefore, this study aims to investigate the feasibility of injecting MagTrace before NACT and then identify the sentinel node at surgery, three to six months later. The aim is also to investigate if a metastatic lymph node can be marked with Magseed® before NACT and together with MagTrace identify the metastatic node, as well as additional sentinel nodes at surgery, three to six months later.

The overall aim is to facilitate logistics at surgery, finding the right SN and minimize axillary surgery.

OBJECTIVES:

Primary objectives:

1. Cohort 1, Node Negative Patients before NACT: To evaluate the SN detection rate with Magtrace® injected before NACT
2. Cohort 2, Node Positive Patients before NACT: To evaluate per-operative identification and removal rate of a Magseed clipped metastatic index lymph node

Secondary objectives:

1. Node Negative Patients before NACT: To evaluate the concordance of SN detection by Magtrace® injected before NACT and Technetium (Tc99) +/- blue dye (BD) injected after NACT, respectively
2. Node Positive Patients before NACT: To evaluate:

   * the SN detection rate with Magtrace® injected before NACT
   * the concordance of SNs detected by Magtrace® injected before NACT and Tc99 + BD injected after NACT, during targeted axillary dissection (TAD)
   * the number of metastatic SNs and metastatic additional lymph nodes from the axillary dissection

ENDPOINTS:

Primary endpoints:

* Cohort 1, SN detection rate
* Cohort 2, Identification rate and removal rate of clipped index metastatic lymph node

Secondary endpoints:

* Cohort 1, Concordance of SNs identified with Magtrace and Tc99 after NACT
* Cohort 2, a) SN detection rate. b) Concordance of SNs identified with MagTrace and Tc99 after NACT. c) Number of metastatic lymph nodes among SNs and additional lymph nodes
* Cohort 1+2, Incidence of serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* A patient meeting the following criteria is eligible for participation in the study:
* Patients 18 years of age or older
* Patients with breast cancer planned to undergo preoperative chemotherapy (NACT) with a) planned sentinel lymph node biopsy (SNB) or b) axillary lymph node dissection, in conjunction with the beast surgery after NACT

Exclusion Criteria:

* Intolerance / hypersensitivity to iron or dextran compounds or SPIO.
* Patients who are required to undergo MR to evaluate tumour response
* Pregnancy or breast feeding
* Patients with an iron overload disease.
* Patient deprived of liberty or under guardianship.
* Inability to understand given information, give informed consent, undergo study procedures
* MRI (subgroup of patients): Conditions contraindicating MRI including, but not limited to, BMI > 40 kg/m2, claustrophobia, metallic implants or internal electrical devices (e.g. Pacemaker).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Detection rate of axillary sentinel node after neoadjuvant chemotherapy | Time between injection of magnetic tracer and technetium-99 is between 3-4 months-
  Cohort 1: Patients with clinically node negative axillary nodes who undergo neoadjuatnt chemotherapy- Injected with Magtrace (magnetic non particles) near the breast cancer. Detection rate of SN using magtrace to be compared with there rate using the standard comparator Technetium-99
Detection rate of pre-marked metastatic axillary node(s) with magseed after neoadjuvant chemotherapy | Time between magseed insertion of magnetic tracer and surgery will be 3-4 months
  Cohort 2: Patients with clinically node positive axillary nodes who undergo neoadjuatnt chemotherapy- Injected with Magtrace (magnetic non particles) near the breast cancer. Detection rate of SN using magtrace to be compared with there rate using the standard comparator Technetium-99

SECONDARY OUTCOMES:
Concordance rate of axillary Sentinel Node (SN) identified with BOTH MagTrace and Technetium-99 after neoadjuvant chemotherapy | Time between injection of magnetic tracer and technetium-99 is between 3-4 months-
  Cohort 1: Lymph nodes removed that contain BOTH Magtrace and Technetium-99
Concordance rate of Sentinel Node and non-Sentinel Nodes identified with BOTH magtrace and technetium-99 | Time between injection of magnetic tracer and technetium-99 is between 3-4 months-
  Cohort 2: Patients with clinically node positive axillary nodes who undergo neoadjuvant chemotherapy. Targeted axillary dissection followed by axillary clearance to be carried out for comparison of concordance rates
Incidence of serious adverse events (SAEs) | Through study completion, an average of 1 year
  For both cohort 1 and 2: clinically node negative and positive patients respectively

CONTACTS AND LOCATIONS:
Overall Officials: Fedrik Warnberg, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher CS, Margenthaler JA, Hunt KK, Schwartz T. The Landmark Series: Axillary Management in Breast Cancer. Ann Surg Oncol. 2020 Mar;27(3):724-729. doi: 10.1245/s10434-019-08154-5. Epub 2019 Dec 20. PMID 31863417
- [Background] Racz JM, Caudle AS. Sentinel Node Lymph Node Surgery After Neoadjuvant Therapy: Principles and Techniques. Ann Surg Oncol. 2019 Oct;26(10):3040-3045. doi: 10.1245/s10434-019-07591-6. Epub 2019 Jul 24. PMID 31342394
- [Background] Samiei S, van Kaathoven BN, Boersma L, Granzier RWY, Siesling S, Engelen SME, de Munck L, van Kuijk SMJ, van der Hulst RRJW, Lobbes MBI, Smidt ML, van Nijnatten TJA. Risk of Positive Sentinel Lymph Node After Neoadjuvant Systemic Therapy in Clinically Node-Negative Breast Cancer: Implications for Postmastectomy Radiation Therapy and Immediate Breast Reconstruction. Ann Surg Oncol. 2019 Nov;26(12):3902-3909. doi: 10.1245/s10434-019-07643-x. Epub 2019 Jul 29. PMID 31359276
- [Background] Warnberg F, Stigberg E, Obondo C, Olofsson H, Abdsaleh S, Warnberg M, Karakatsanis A. Long-Term Outcome After Retro-Areolar Versus Peri-Tumoral Injection of Superparamagnetic Iron Oxide Nanoparticles (SPIO) for Sentinel Lymph Node Detection in Breast Cancer Surgery. Ann Surg Oncol. 2019 May;26(5):1247-1253. doi: 10.1245/s10434-019-07239-5. Epub 2019 Mar 4. PMID 30830536
- [Background] Karakatsanis A, Hersi AF, Pistiolis L, Olofsson Bagge R, Lykoudis PM, Eriksson S, Warnberg F; SentiNot Trialists Group. Effect of preoperative injection of superparamagnetic iron oxide particles on rates of sentinel lymph node dissection in women undergoing surgery for ductal carcinoma in situ (SentiNot study). Br J Surg. 2019 May;106(6):720-728. doi: 10.1002/bjs.11110. Epub 2019 Mar 6. PMID 30839104
- [Background] Brown AS, Hunt KK, Shen J, Huo L, Babiera GV, Ross MI, Meric-Bernstam F, Feig BW, Kuerer HM, Boughey JC, Ching CD, Gilcrease MZ. Histologic changes associated with false-negative sentinel lymph nodes after preoperative chemotherapy in patients with confirmed lymph node-positive breast cancer before treatment. Cancer. 2010 Jun 15;116(12):2878-83. doi: 10.1002/cncr.25066. PMID 20564394
- [Background] Greenwood HI, Wong JM, Mukhtar RA, Alvarado MD, Price ER. Feasibility of Magnetic Seeds for Preoperative Localization of Axillary Lymph Nodes in Breast Cancer Treatment. AJR Am J Roentgenol. 2019 Oct;213(4):953-957. doi: 10.2214/AJR.19.21378. Epub 2019 Jun 5. PMID 31166765